CLINICAL TRIAL: NCT03903913
Title: A Phase IIa Open Label Study to Evaluate the Safety, Tolerability and Efficacy of S-1226 Administered by Nebulization in Subjects With Mild to Moderate Cystic Fibrosis and Non CF Bronchiectasis
Brief Title: Safety, Tolerability and Efficacy of S-1226 in Cystic Fibrosis and Non CF Bronchiectasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SolAeroMed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SAMi-03-1-01
Record Dates: First submitted 2019-02-15; First posted 2019-04-04 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Cystic Fibrosis; Bronchiectasis
Keywords: Asthma; Carbon dioxide; Perfluorocarbon; Mucolytic
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis; Asthma | interventions — perfluorooctylbromide and CO2 drug combination

STUDY DESIGN:
Intervention Model Description: Single center, open label, Phase IIa, sequential, multiple-ascending dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Study (Experimental): Subjects will receive up to three inhaled doses of S- 1226. Each dose will be administered over a 2-minute treatment period (with a minimum 2-minute break between treatments) with a nebulizer as follows.
  Three S-1226 formulations will be tested sequentially:
  * S-1226(4%) is composed of 3 mL PFOB and 4% CO2
  * S-1226(8%) is composed of 3 mL PFOB and 8% CO2
  * S-1226(12%) is composed of 3 mL PFOB and 12% CO2
  Each formulation will be administered by inhalation for a period of 2 minutes.The nebulizer will be filled with 3 mL of PFOB. The nebulizer is connected to a compressed medical gas mixture consisting of either 4%, 8% or 12%, CO2. A driving pressure of 20 psi will be used, producing a gas flow rate of 9 L/min.
  Interventions: Drug: S-1226
- Daily Dosing Study (Experimental): Eligible subjects will receive S-1226 twice daily for 5 consecutive days. Subjects will receive up to three doses of S-1226 in the morning and afternoon, administered over three 2-minute periods with a Circulaire nebulizer, filled with one of the dosages outlined below, depending on the safety and tolerability data gathered from the dose escalation study for that particular subject.
  * S-1226(4%) is composed of 3 mL PFOB and 4% CO2
  * S-1226(8%) is composed of 3 mL PFOB and 8% CO2
  * S-1226(12%) is composed of 3 mL PFOB and 12% CO2
  Interventions: Drug: S-1226

INTERVENTIONS:
Drug: S-1226 — The drug product S-1226 has two components delivered by inhalation. It is a mixture of perfluorooctylbromide (PFOB) nebulized with a medical gas mixture containing CO2. The PFOB component remains the same but the medical gas component contains 4%, 8% or 12% CO2.
  Other Names: S-1226 (4%); S-1226 (8%); S-1226 (12%)

SUMMARY:
This is a single center, open label, Phase IIa, multiple-ascending dose study in which subjects with mild to moderate Cystic Fibrosis and non CF bronchiectasis (n≤12) will be enrolled.

The safety and tolerability of S-1226 composed of PFOB with ascending doses of carbon dioxide (4%, 8%, and 12% CO2) administered twice daily in subjects with Cystic Fibrosis and non CF bronchiectasis will be evaluated. This will be followed by 5 day consecutive treatment using the highest tolerated dose of S1226. Participants can choose additional use of a further four weeks (28 days) of S-1226 therapy at home, using same or a lower tolerated dose.

DETAILED DESCRIPTION:
This is a single center, open label, Phase IIa, multiple-ascending dose study in which subjects with mild to moderate Cystic Fibrosis and non CF bronchiectasis (n≤12) will be enrolled.

The study will consist of a screening period, a run-in and two dosing and evaluation periods (with a minimum two-day break in between) and a follow-up period.

The dosing and evaluation period of the study is divided into two consecutive components:

1. Dose escalation study

   - This segment of the treatment period is designed to assess the safety and tolerability of escalating doses of S-1226 (4%, 8% and 12%) in those with mild-moderate CF and non CF bronchiectasis
2. Daily dosing study - This segment of the treatment period is designed to assess the short term (5 day) safety and tolerability of twice daily administration of a fixed dose of S-1226 in subjects with mild-moderate CF and non CF bronchiectasis.

The primary aim of this study of S-1226 is to capture information to inform follow-up S-1226 clinical studies in CF and non CF bronchiectasis. Important in this regard will be data on safety, tolerability, dosing and efficacy. Specifically, regarding efficacy, the investigators want to examine for optimal dose ranging and magnitude of the effect to determine the power calculations for any follow-up studies and to determine which outcome measures best reflect the effects of the drug. Because the study is investigational in nature, it will be un-blinded and information will be analyzed as it is collected.

During the screening and the run-in period, the subjects will have safety assessments and all eligibility criteria confirmed. The run-in period involves meeting with the study subjects 1 - 2 weeks prior to the start of the treatment for a physical exam, concomitant medication review, spirometry and information regarding the study. The consent process will also take place at this stage.

The dose escalation period will include 3 days of twice daily treatment of the study drug with a washout period in between. The dose of CO2 in S-1226 will be sequentially escalated for the particular subject from the starting dose of 4% CO2. Planned subsequent dose levels are 8% and 12% CO2, although doses may be adjusted within this range based on safety and tolerability data from the completed dosing days. Subjects will not be dosed with a higher CO2 level until drug administration of the preceding dose level has been completed and safety data reviewed by the Safety Committee and a decision taken to proceed or not with the next sequential dose level.

There will be a washout period between the dose escalation and the daily dosing study. The daily dosing study will include 5 days of twice daily treatment of the study drug based on the results of the dose escalation study. Lung function tests will be performed before and after the treatment.

Subjects in the Home Extension Study will receive S-1226 twice daily for 28 consecutive days. Subjects will monitor daily symptom scores. Oxygen saturation values, as determined by pulse oximetry, will be monitored 2 minutes prior to therapy, during therapy and for up to 30 minutes post therapy. Pulmonary function studies will be assessed weekly by the designated respiratory therapist between 4-7 pm.

The follow-up phase will occur 10-14 days after completion of the final dose. This will involve a clinical exam, spirometry and completion of CFQ-R.

ELIGIBILITY:
Inclusion Criterian(CF lung disease):

* Confirmed diagnosis of Cystic Fibrosis by sweat chloride concentration over 60 mosm/L and/or genotype analysis identifying two disease causing mutations
* Male or Female over the age of 14
* Followed in CF clinic at Foothills Hospital or Alberta Children's Hospital
* Known lung involvement

  1. Recommended airway clearance daily or twice daily
  2. FEV1, % predicted, between 40-80%
  3. Evidence of Cystic Fibrosis lung involvement on Imaging, if available
* Competent at providing reliable and accurate pulmonary function studies
* Clinically stable - no pulmonary exacerbation of CF for which the patient has been hospitalized or received intravenous antibiotics for 4 weeks, no change in frequency of airway clearance

Exclusion Criteria CF lung disease:

* Gross Hemoptysis in previous 4 weeks
* Pneumothorax in previous 4 weeks
* Pregnancy or of child bearing age without adequate contraception
* Inability to produce acceptable and reproducible pulmonary function studies
* Evidence of elevated PaCO2 in recent 6 months
* Inability to perform airway clearance twice a day for the duration of the study
* History of anxiety/panic disorders
* Breast-feeding subject.
* Positive pregnancy test at screening.
* Subject, who in the opinion of the Investigator, is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.

Gross Hemoptysis in previous 4 weeks Pneumothorax in previous 4 weeks Pregnancy or of child bearing age without adequate contraception Inability to produce acceptable and reproducible pulmonary function studies Evidence of elevated PaCO2 in recent 6 months Inability to perform airway clearance twice a day for the duration of the study History of anxiety/panic disorders Breast-feeding subject. Positive pregnancy test at screening. Subject, who in the opinion of the Investigator, is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.

Inclusion Criteria (Non-CF bronchiectasis)

* Male or Female including and over the age of 14
* Known lung involvement

  1. FEV1, % predicted, between 40-80%
  2. Evidence of bronchiectasis on Imaging
* Competent at providing reliable and accurate pulmonary function studies
* Clinically stable - no pulmonary exacerbation for which the patient has been hospitalized or received intravenous antibiotics for 4 weeks

Exclusion Criteria (Non-CF bronchiectasis)

* Diagnosis of Cystic Fibrosis
* Active tuberculosis and/or non-tuberculosis mycobacterial infection
* Active allergic bronchopulmonary aspergillosis
* Traction bronchiectasis due to pulmonary fibrosis
* Gross Hemoptysis in previous 4 weeks
* Pneumothorax in previous 4 weeks
* Pregnancy or of child bearing age without adequate contraception
* Inability to produce acceptable and reproducible pulmonary function studies
* Evidence of elevated PaCO2 in recent 6 months
* Inability to perform airway clearance twice a day for the duration of the study
* History of anxiety/panic disorders
* Breast-feeding subject.
* Positive pregnancy test at screening.
* Subject, who in the opinion of the Investigator, is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | 60 minutes
  The number and percent of treatment emergent adverse events will be monitored, recorded and graded for severity and assigned attribution. The severity will be assessed in the following manner:
  Mild: Awareness of signs or symptoms, but are easily tolerated and are of minor irritant type, causing no limitations of usual activities. Signs or symptoms may require minor action or additional therapy.
  Moderate: Discomfort severe enough to cause some limitations of usual activities and may require action or additional therapy.
  Severe: Incapacitating with inability to carry out usual activities and requires specific action and/or medical attention. Note: the term severe is not the same as "serious", which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

SECONDARY OUTCOMES:
Change from baseline in percent of predicted forced expiratory volume in 1 Second | 60 minutes
  Change from baseline in percent of predicted forced expiratory volume in 1 Second (FEV1) will be calculated by measuring FEV1 at baseline and after treatment. FEV1 is defined as the volume of air exhaled from the lungs in the first second of a forced expiration.
Change from baseline in the respiratory domain of Cystic Fibrosis Questionnaire -Revised | Up to 4 weeks
  Change from baseline in respiratory symptoms scores (subscale) of the Cystic Fibrosis Questionnaire -Revised (CFQ-R) will be measured. CFQ-R is a validated, disease specific, patient reported outcome measure used to evaluate the impact of CF on overall health, daily life, and perceived well-being and symptoms. This sub-scale ranges from scores of 0-100, with higher values representing a better outcome.

OTHER OUTCOMES:
Change from baseline in Forced Vital Capacity | Up to 4 weeks
  Change from baseline in Forced Vital Capacity (FVC) will be measured. FVC is the total volume of air that can be exhaled during a maximal forced expiration effort.
Change from baseline in Forced Expiratory Flow at 25-75% | Up to 4 weeks
  Change from baseline in Forced Expiratory Flow at 25-75% (FEF25-75%) will be measured. FEF25-75% is defined as Forced expiratory flow over the middle one half of the Forced Vital Capacity (FVC); the average flow from the point at which 25 percent of the FVC has been exhaled to the point at which 75 percent of the FVC has been exhaled.
Change from baseline in Inspiratory Capacity | Up to 4 weeks
  Change from baseline in Inspiratory Capacity (IC) will be measured. IC is defined as the maximal volume of air that can be inhaled from the resting expiratory level.
Change from baseline in Thoracic Gas Volume | Up to 4 weeks
  Change from baseline in Thoracic Gas Volume (TGV) will be measured. TGV is defined as the absolute volume of gas in the thorax at any point in time and any level of alveolar pressure.
Change from baseline in Residual Volume | Up to 4 weeks
  Change from baseline in Residual Volume (RV) will be measured. RV is defined as the volume of air remaining in the lungs after a maximal exhalation.
Change from baseline in Lung Clearance Index | Up to 4 weeks
  Change from baseline in Lung Clearance Index will be measured. Lung clearance index is a unitless measurement, which is defined as the total volume of expired gas required to decrease the amount of the tracer gas to 1/40 of its initial concentration divided by the functional residual capacity. It is measure of ventilation inhomogeneity.
Change in expectorated sputum volume | 120 minutes
  Expectorated sputum volume (in milliliters) will be measured at baseline and after treatment and any changes in measured volume from baseline will be reported.
Change from baseline in oxygen saturation | 60 minutes
  Change from baseline in percent of oxygen saturation (measured by pulse oximetry) will be calculated by measuring oxygen saturation before and up to 60 minutes after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Montgomery, MD, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Adult Cystic Fibrosis Clinic at the Foothills Hospital, Calgary, Alberta
  - Pediatric Cystic Fibrosis Clinic at Alberta Children's Hospital, Calgary, Alberta
  - Alberta Lung Function, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swystun V, Green FHY, Dennis JH, Rampakakis E, Lalli G, Fadayomi M, Chiu A, Shrestha G, El Shahat SG, Nelson DE, El Mays TY, Pieron CA, Leigh R. A phase IIa proof-of-concept, placebo-controlled, randomized, double-blind, crossover, single-dose clinical trial of a new class of bronchodilator for acute asthma. Trials. 2018 Jun 18;19(1):321. doi: 10.1186/s13063-018-2720-6. PMID 29914544
- [Background] Green FH, Leigh R, Fadayomi M, Lalli G, Chiu A, Shrestha G, ElShahat SG, Nelson DE, El Mays TY, Pieron CA, Dennis JH. A phase I, placebo-controlled, randomized, double-blind, single ascending dose-ranging study to evaluate the safety and tolerability of a novel biophysical bronchodilator (S-1226) administered by nebulization in healthy volunteers. Trials. 2016 Jul 28;17:361. doi: 10.1186/s13063-016-1489-8. PMID 27464582
- [Background] El Mays TY, Choudhury P, Leigh R, Koumoundouros E, Van der Velden J, Shrestha G, Pieron CA, Dennis JH, Green FH, Snibson KJ. Nebulized perflubron and carbon dioxide rapidly dilate constricted airways in an ovine model of allergic asthma. Respir Res. 2014 Sep 16;15(1):98. doi: 10.1186/s12931-014-0098-x. PMID 25355286